CLINICAL TRIAL: NCT04376554
Title: Phase 1 Study to Evaluate the Effect of Oral Administration of Tebipenem Pivoxil Hydrobromide on Normal Human Intestinal Microbiota in Healthy Volunteers
Brief Title: Effect of Tebipenem on Normal Human Intestinal Microbiota
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Spero Therapeutics (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPR994-103
Record Dates: First submitted 2020-03-16; First posted 2020-05-06 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Healthy Volunteers
Keywords: intestinal microbiota; safety; pharmacokinetics; TBPM-PI-HBr; tebipenem
MeSH Terms: interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Intervention Model Description: Single-Center, Open-Label, Randomized, Parallel-Group, Active Control, Phase 1 Study
Masking Description: Subjects will be randomized by gender to 1:1 ratio to receive TBPM-PI-HBr or amoxicillin-clavulanate using a SAS ® generated randomization code and the treatment allocation will be performed using a block randomization algorithm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TBPM-PI-HBr (Experimental): Healthy subjects meeting eligibility criteria will be sequentially randomized to receive either 600mg TBPM-PI-HBr every 8 hours (PO q8h [±1 hour]) or 500/125mg amoxicillin-clavulanate PO q8h (±1 hour) for 10 days.
  Interventions: Drug: TBPM-PI-HBr
- amoxicillin-clavulanate (Active Comparator): Healthy subjects meeting eligibility criteria will be sequentially randomized to receive either 500/125mg amoxicillin-clavulanate PO q8h (±1 hour) or 600mg TBPM-PI-HBr every 8 hours (PO q8h [±1 hour]) or for 10 days.
  Interventions: Drug: amoxicillin-clavulanate

INTERVENTIONS:
Drug: TBPM-PI-HBr — TBPM-PI-HBr (2 x 300mg tablets) PO q8h [±1 hour] for 10 days
  Other Names: TBPM-PI-HBr oral tablet
  Arms: TBPM-PI-HBr
Drug: amoxicillin-clavulanate — amoxicillin-clavulanate (1 × 500mg/125mg tablet) PO q8h [±1 hour] for 10 days
  Other Names: amoxicillin-clavulanate oral tablets
  Arms: amoxicillin-clavulanate

SUMMARY:
The overall purpose of this study is to support the development of an oral formulation of TBPM-PI-HBr by assessing the potential ecological effects of tebipenem on the normal intestinal microbiota as compared to the effects of oral amoxicillin-clavulanate.

DETAILED DESCRIPTION:
This is a single-center, open-label, randomized, parallel-group, active-control, phase 1 study consisting of 10-day treatment period using TBPM-PI-HBr (600mg) (2× 300mg film coated tablets) or amoxicillin-clavulanate (500mg/125mg) orally every 8 hours (PO q8h [±1 hour]) in healthy volunteers. Participants will be randomized by gender to 1:1 ratio on Day 1. A maximum of 30 participants will be randomly assigned to the study treatment groups (15 in each arm) such that approximately 24 evaluable participants complete the study. Due to the multidimensional nature of data of the study, a power statement on a single endpoint is not appropriate. The main aim of the study is to estimate the effects of treatment on the intestinal microbiota, and to assess the pattern of susceptibility to specific pathogens. Based upon previous studies, a sample size of 12 participants in each group is considered sufficient to demonstrate a clinically significant impact of antibiotics on the microbiota. Total duration of study participation for each participant will be approximately 7 months.Screening visit will be performed between Day -28 to Day -1. Randomization will be performed on Day 1 and with treatment being administered from Day 1 to Day 10. Follow-up of participants will occur on Day 14, 21, 90 and 180 with appropriate visit windows. Adverse events and concomitant medications will be recorded until the end of the study (Day 180).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult males and/or females, ≥18 years of age at the time of screening;
2. Medically healthy without clinically significant abnormal values for hematology, clinical chemistry, urinalysis, physical examination, vital signs, or ECG as determined by the investigator during the screening period. Discussion is encouraged between the Investigator and the Sponsor Medical Monitor regarding the clinical relevance of any abnormal laboratory value during the pre-dose period;
3. Willing and able to provide written informed consent;
4. Willing and able to comply with all study assessments and adhere to the protocol schedule, including all scheduled post-therapy visits;
5. Have suitable venous access for blood sampling;
6. Women of childbearing potential (WOCBP*) must use a highly effective form of birth control (confirmed by the Investigator). Rhythm methods will not be considered as highly effective methods of birth control. WOCBP must agree to use a highly effective method of birth control, as defined above, from signing the Informed Consent Form (ICF), throughout the study duration and until 30 days after the last dose of study drug;
7. Non-vasectomized male volunteers must use an adequate method of contraception (condom or condom with spermicide, depending on local regulations) from the time of signing the ICF, throughout the study duration and until 30 days after the last dose of study drug. Men with a partner who is (are) not of childbearing potential are exempt from these requirements;
8. Male volunteers must not donate sperm for time of signing the ICF until at least 30 days after the last dose of the study drug

Exclusion Criteria:

1. History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, endocrine, immunologic, dermatologic or neurological disease, including any acute illness or surgery within the past 3 months determined by the Investigator to be clinically relevant;
2. History or presence of known or suspected gastrointestinal disorder, including but not limited to Clostridioides difficile infection, inflammatory bowel disease, recent history of food poisoning or other stomach/intestinal disorders including gastroenteritis (within 6 months);
3. History of systemic antibiotic treatment during the last three months prior to randomization;
4. Use of any systemic prescription medication or any systemic over-the-counter medication, including herbal products and vitamins or probiotics within 7 days prior to randomization; except for hormonal contraceptives and the intermittent use of paracetamol, ibuprofen, and antihistamines;
5. Alanine transaminase (ALT) or aspartate transaminase (AST) >5 × upper limit of normal and CrCl of ≤50 mL/min, as estimated by the Lund-Malmö revised formula;
6. History of seizure disorders, except for febrile seizures in childhood;
7. History of substance or alcohol abuse and positive urine drug testing at screening. History of substance or alcohol abuse and negative urine drug testing at screening can be enrolled in study based on the Investigator's discretion;
8. Positive for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (HCV);
9. Documented or suspected hypersensitivity reaction or anaphylaxis to β-lactam antibiotics (e.g., cephalosporins, penicillins, carbapenems), product excipients (Mannitol, microcrystalline cellulose, crospovidone, magnesium stearate, colloidal silicon dioxide, and film coating systems [Opadry]) or any contraindication to the use of amoxicillin- clavulanate;
10. Participation in another investigational clinical study within 3 months prior to Day 1;
11. Current or anticipated need for systemic antibiotics, probiotics, or laxatives during the study;
12. Any other condition or prior therapy, which, in the opinion of the Investigator, would make the volunteer unsuitable for this study, including inability to cooperate fully with the requirements of the study protocol or likely to be non-compliant with any study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2021-04-06 (Actual); Study Completion 2021-04-06 (Actual)

PRIMARY OUTCOMES:
Changes in the number of microorganisms in the intestinal flora of healthy subjects during and after 10 days of oral administration of TBPM-PI-HBr or amoxicillin-clavulanate | Change from baseline (Day-1), at Days 2, 4, 7, 10, 14, 21, 90, and 180
  Changes in the number of microorganisms identified in feces
Changes in the types of microorganisms in the intestinal flora of healthy subjects during and after 10 days of oral administration of TBPM-PI-HBr or amoxicillin-clavulanate | Change from baseline (Day-1), at Days 2, 4, 7, 10, 14, 21, 90, and 180
  Changes in the types of microorganisms identified in feces

SECONDARY OUTCOMES:
To explore the potential for development of resistance by measuring the number of new colonizing bacterial isolates | Change from baseline (Day-1), at Days 2, 4, 7, 10, 14, 21, 90, and 180
  Emergence of resistant strains with increasing minimum inhibitory concentration values during treatment and post-treatment with tebipenem and amoxicillin-clavulanate will be determined from fecal samples.
To assess the plasma concentrations of tebipenem over 10 days of oral administration of TBPM-PI-HBr. | Day 1 through Day 14
  PK concentration of tebipenem will be measured in plasma. Concentrations of tebipenem will be plotted for each participant.
To assess the fecal concentrations of tebipenem over 10 days of oral administration of TBPM-PI-HBr. | Day 1 through Day 14
  PK concentration of tebipenem will be measured in feces.Concentrations of tebipenem will be plotted for each participant.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Incidents of treatment-emergent adverse events from Day 1 through last follow-up visit (180 days after last dose)
  To assess the incidents of treatment-emergent adverse events following 10 days of oral TBPM-PI-HBr administration
Incidence of abnormal safety laboratory assessments [Safety and Tolerability] | Incidents of abnormal safety laboratory assessments from Day 1 through last follow-up visit (180 days after last dose)
  To assess the incidents of abnormal hematology, biochemistry, coagulation and urinalysis assessments following 10 days of oral TBPM-PI-HBr administration
Incidence of abnormal vital sign assessments [Safety and Tolerability] | Incidents of abnormal vital sign assessments from Day 1 through last follow-up visit (180 days after last dose)
  To assess the incidents of abnormal heart rate, blood pressure and body temperature assessments following 10 days of oral TBPM-PI-HBr administration
Incidence of abnormal physical exam assessments [Safety and Tolerability] | Incidents of abnormal physical exam assessments from Day 1 through last follow-up visit (180 days after last dose)
  To assess the incidents of abnormal body system assessments following 10 days of oral TBPM-PI-HBr administration

OTHER OUTCOMES:
Correlation of intestinal microbiota patterns with tebipenem concentrations measured in feces. | Day 1 through last follow-up visit (180 days after last dose)
  Measurement of concentrations of TBPM in feces using bioactivity techniques and correlate changes in microbiota as evidenced by various microbiological techniques (eg. microbial diversity, colony counts, and molecular methods).

CONTACTS AND LOCATIONS:
Overall Officials: Steffan Rosenborg, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Huddinge, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sewunet T, Razavi M, Rosenborg S, Camporeale A, Nowak M, Melnick D, Gasink LB, Eckburg PB, Critchley IA, Nord CE, Giske CG. Effect of tebipenem pivoxil hydrobromide on the normal gut microbiota of a healthy adult population in Sweden: a randomised controlled trial. Lancet Microbe. 2024 Apr;5(4):e355-e365. doi: 10.1016/S2666-5247(23)00360-9. Epub 2024 Feb 29. PMID 38432233